CLINICAL TRIAL: NCT01430208
Title: New Mini-resectoscope as Alternative to Traditional Hysteroscopy in the Treatment of Uterine Lesions
Brief Title: A New Alternative to Traditional Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Maurizio Guido, medical doctor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUMREP-11-0778
Record Dates: First submitted 2011-09-02; First posted 2011-09-08 (Estimated); Last update posted 2011-09-08 (Estimated); Status verified 2011-09

CONDITIONS: Intrauterine Diseases; Myomas; Polyps
Keywords: endometrial pathology
MeSH Terms: conditions — Myoma; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- mini-resectoscope (Active Comparator)
  Interventions: Procedure: resectoscopy
- tradiorional resectoscope (Active Comparator)
  Interventions: Procedure: resectoscopy
- bettocchi resectoscope (Active Comparator)
  Interventions: Procedure: resectoscopy

INTERVENTIONS:
Procedure: resectoscopy — hysteroscopy for myomas G0 and/or polyps

SUMMARY:
Hysteroscopy is a procedure designed for the diagnosis and the treatment of intra-uterine diseases. The development of smaller hysteroscopes allowed to change the approach to the intra-uterine lesions unifying the diagnostic and operative time. Recently Gubbini et al. developed a mini-resectoscope feasible for "see&treat" hysteroscopy. The objective of the study is to compare the new 16 Fr mini28 resectoscope by Gubbini with Traditional 22 Fr resectoscope and Bettocchi 15 Fr hysteroscope for the treatment of uterine cavitary lesions. The investigators enrolled 401 women affected by endometrial polyps and/or G0 myomas, randomly allocated to receive the treatment with traditional resectoscope (127 women), with mini-resectoscope by Gubbini (142 women) and Bettocchi hysteroscope (132 women). Operating time, distension media delivered, dismiss time and discomfort experienced were recorded.

ELIGIBILITY:
Inclusion Criteria:

* women between 18-75 years of age
* endometrial polyps and/or G0 myomas smaller than 3 cm of diameter

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2010-01; Primary Completion 2011-04 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
efficacy of the treatment with mini-resectoscope in comparison with the traditional hysteroscopy in the whole group of 401 patients | sixteen months
  Operating time (min), distension media used (ml), dismiss time (hours), patients discomfort (VAS)

SECONDARY OUTCOMES:
efficacy of the treatment with mini-resectoscope in comparison with the traditional hysteroscopy in the treatment of intrauterine lesions larger than 1,5cm in diameter | sixteen months
  Operating time(min), distension media used (ml), dismiss time (hours), patients discomfort (VAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic university of Sacred Heart, Rome, Rome, Italy

REFERENCES:
- [Derived] Ricciardi R, Lanzone A, Tagliaferri V, Di Florio C, Ricciardi L, Selvaggi L, Guido M. Using a 16-French resectoscope as an alternative device in the treatment of uterine lesions: a randomized controlled trial. Obstet Gynecol. 2012 Jul;120(1):160-5. doi: 10.1097/AOG.0b013e31825b9086. PMID 22914405